CLINICAL TRIAL: NCT04074395
Title: A Retrospective Analysis of Oral and Maxillofacial Pathological Lesions in Egyptian Children
Brief Title: Oral and Maxillofacial Pathology in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Mohsen Aly, lecturer in pediatric dentistry and dental public health, faculty of dentistry, Cairo university, Cairo University
Other Study IDs: Oral pathology
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Mouth Diseases
Keywords: oral pathology
MeSH Terms: conditions — Mouth Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
determination of the relative frequency of oral and maxillofacial pathological lesions among the Egyptian children and compare it with the global reports.

DETAILED DESCRIPTION:
Oral and maxillofacial pathology in pediatric patients differs from the general population, as the nature of lesions in children changes with growth and development. Oral and maxillofacial pathology encompasses a wide spectrum of diseases, some of which (i.e. aphthous ulceration, geographic tongue, and herpes labialis) can be diagnosed on clinical presentation alone. For other soft tissue diseases and for pathology with bony components, incisional or excisional biopsy is mandatory to establish a definitive diagnosis .

Several studies illustrated that oral and maxillofacial pathology in pediatric populations varies based on the geographic location of the population as racial and environmental specificities and the lifestyle of each population may influence the prevalence of these diseases .

Although there is increasing literature regarding the incidence and prevalence of pediatric oral and maxillofacial pathology, there is no study investigating the range and frequency in Egyptian children.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy records for children aged from 0 to 18 years

Exclusion Criteria:

* Biopsy records for patients older than 18
* Incomplete record regarding age, gender, location

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Biopsy records for children aged from 0 to 18 years
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Frequency of oral and maxillofacial pathological lesions among Egyptian children | one month
  percentage of cases with oral pathological lesions

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt